CLINICAL TRIAL: NCT02955680
Title: Comparison Between Recorded Mother's and Stranger's Voice on the Emergence of General Anesthesia on Pediatric Patients
Brief Title: Recorded Maternal Voice on the Emergence of General Anesthesia on Pediatric Patients
Acronym: Maternal voice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daegu Catholic University Medical Center (Other)
Responsible Party: Principal Investigator, Eugene Kim, Assistant professor, Daegu Catholic University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: DCUMC_2
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Anesthesia, General
Keywords: emergence delirium; emergence time; bispectral index
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Group M (Experimental): At the end of surgery, patients were stimulated to wake up by recorded mother's voice, which was recorded before the operation.
  Interventions: Procedure: recorded maternal voice
- Group S (Active Comparator): At the end of surgery, patients were stimulated to wake up by recorded stranger's voice, which was recorded before the operation.
  Interventions: Procedure: recorded stranger's voice

INTERVENTIONS:
Procedure: recorded maternal voice — A voice recording will be performed before the operation. At a preoperative visit or preoperative clinic, informed consent was obtained before the recording. On a calm environment, the mother was asked to speak following sentences.
  " OO (first name of child), wake up~. Let's go home with mommy. OO, wake up~. Open your eyes. Take a deep breath. " At the end of surgery, the recorded maternal voice was delivered to the child every 15 seconds until he/she wakes up.
  Arms: Group M
Procedure: recorded stranger's voice — A voice recording will be performed before the operation. On a calm environment, a blinded female investigator was asked to speak following sentences.
  " OO (first name of child), wake up~. Let's go home with mommy. OO, wake up~. Open your eyes. Take a deep breath. "
  Arms: Group S

SUMMARY:
Mother spend a large amount of time with their children. It is assumed that mother contributes to their neurological development not only with visual stimuli, but also with auditory stimuli. A recent study revealed that prefrontal cortex can be activated in response to the self-name being spoken by the mother than by a stranger. Therefore, investigators suppose that recorded maternal voice can stimulate the pediatric patients and thereby fasten the emergence from general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 2 and 8 years of American Society of Anesthesiologists physical status (ASA PS) I or II who are planned to receive ophthalmology or otorhinolaryngology surgery under general anesthesia

Exclusion Criteria:

* ASA PS III or IV
* with developmental delay or neurological diseases associated with symptoms of agitation
* refusal of consent
* maternal mutism
* absence of mother
* with allergy or contraindication to use of ketamine (increased intracranial pressure, open-globe injury, and a psychiatric or seizure disorder)

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2016-11; Primary Completion 2017-09 (Actual); Study Completion 2017-09-21 (Actual)

PRIMARY OUTCOMES:
initial PAED score | During 1 minutes after PACU admission
  On arrival at post-anesthesia care unit (PACU), patients were checked PAED. The PAED scale is a validated observational measure of 5 aspects of child behavior (caregiver eye contact, purposeful movement, evidence of awareness of surroundings, restlessness, and inconsolability). Ratings are summed to produce a total score ranging from 0 to 20; greater scores indicate greater severity.

SECONDARY OUTCOMES:
BIS over 60 | During 1 hour after operation
  At the end of operation, investigators stop the anesthetics and carefully watch the bispectral index (BIS) monitor. Simultaneously, investigators check the duration of time from discontinuation of anesthetics until the BIS >60.
Incidence of emergence delirium (ED) | During 60 minutes after PACU admission
  The incidence of emergence delirium (ED) was defined as pediatric anesthesia emergence delirium (PAED) score of >12 or Watcha scale over 3 at PACU.
PAED score on 10, 20, and 30 min | During 60 minutes after PACU admission
  On arrival at post-anesthesia care unit (PACU), patients were checked PAED. The PAED scale is a validated observational measure of 5 aspects of child behavior (caregiver eye contact, purposeful movement, evidence of awareness of surroundings, restlessness, and inconsolability). Ratings are summed to produce a total score ranging from 0 to 20; greater scores indicate greater severity.
Watcha scale on initial, 10, 20, and 30 min | During 60 minutes after PACU admission
  On arrival and 10, 20, and 30 min after PACU admission, patients were checked Watcha scale as following 4-point scale
  1. calm
  2. crying, but can be consoled
  3. Crying, cannot be consoled
  4. Agitated and thrashing around
BIS over 70 and 80 time | During 1 hour after operation
  At the end of operation, investigators stop the anesthetics and carefully watch the bispectral index (BIS) monitor. Simultaneously, investigators check the duration of time from discontinuation of anesthetics until the BIS reached 70 and 80 value.
FLACC score on initial, 10, 20, and 30 min | During 60 minutes after PACU admission
  Face, legs, activity, cry, and consolability (FLACC) score is checked every 10min after PACU admission
Extubation time | During 1 hour after operation
  time from discontinuation of anesthetics to extubation
mean blood pressure | During 1 hour after operation
  Mean blood pressure (MBP) is checked at five time points; cessation of anesthetics (baseline), the BIS reached value of 60, time of extubation, PACU arrival, and PACU discharge.
Heart rate | During 1 hour after operation
  Heart rate is checked at five time points; cessation of anesthetics (baseline), the BIS reached value of 60, time of extubation, PACU arrival, and PACU discharge.
Eye opening or purposeful movement time | During 1 hour after operation
  defined as the interval from the cessation of anesthetics to eye opening or purposeful movement of patients

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Kim, MD, Study Director — Daegu Catholic University Medical Center
Locations (1):
- Daegu Catholic University Medical Center, Daegu, South Korea

REFERENCES:
- [Derived] Byun S, Song S, Kim JH, Ryu T, Jeong MY, Kim E. Mother's recorded voice on emergence can decrease postoperative emergence delirium from general anaesthesia in paediatric patients: a prospective randomised controlled trial. Br J Anaesth. 2018 Aug;121(2):483-489. doi: 10.1016/j.bja.2018.01.042. Epub 2018 Apr 17. PMID 30032889
- [Derived] Song SY, Kwak SG, Kim E. Effect of a mother's recorded voice on emergence from general anesthesia in pediatric patients: study protocol for a randomized controlled trial. Trials. 2017 Sep 15;18(1):430. doi: 10.1186/s13063-017-2164-4. PMID 28915907